CLINICAL TRIAL: NCT04628923
Title: Tthe Anaesthetic Efficacy of Quadratus Lumborum Block by Paraspinous Sagittal Shift Approach for Hip Surgery:a Case Series
Brief Title: Quadratus Lumborum Block by Paraspinous Sagittal Shift Approach for Hip Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, Assistant professor Doaa Rashwan, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FMBSUREC/05072020/AbdEl Badei2
Record Dates: First submitted 2020-09-18; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Self Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLB (Experimental): With the patient in the lateral decubitus and the block side independent, a curvilinear ultrasound transducer (2-5 MHz) will be directed caudally in a sagittal plane 3-4 cm lateral to the lumbar spinous process of L4, which is almost opposite to the iliac crest, producing a longitudinal scan of the lumbar paravertebral region; and thus identifying the transverse processes of L3 and L4, with PM muscle in-between and erector spinae muscle posteriorly.
  The probe is shifted slowly to the lateral side until the transverse processes disappear and the QL muscle is evident in its long axis attached caudally to the iliac crest with a characteristic sonographic image of three muscle layers appearing from posterior to anterior as: erector spinae, QL, and PM muscles respectively.
  Interventions: Other: QUADRATUS LUMBORUM BLOCK

INTERVENTIONS:
Other: QUADRATUS LUMBORUM BLOCK — QUADRATUS LUMBORUM BLOCK BY PARASPINOUS SAGITTAL SHIFT APPROACH

SUMMARY:
The quadratus lumborum block (QLB) was first described by Blanco. it is a compartment block procedure during which a local anesthetic is injected into the muscle plane of the quadratus lumborum (QL) muscle under ultrasound guidance Currently, QLB is divided into four types based on the injection point of the local anesthetic: lateral, anterior, posterior, and intramuscular QLB. QLB is widely used for various types of abdominal surgeries (

DETAILED DESCRIPTION:
the investigators will evaluate the anesthetic efficacy of quadratus lumborum block by paraspinous sagittal shift approach for hip surgery by injecting 30 ml of 0. 5% bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

-ASA I and II

Exclusion Criteria:

* Contraindications for regional blocks (eg. Patient refusal Infection at the injection site, coagulopathy)
* Allergic reaction to drugs.
* opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
sensory and motor block level | immediately after the intervention/procedure/surgery
  BY PIN PRICK

IPD SHARING:
Plan to Share IPD: No